CLINICAL TRIAL: NCT04875884
Title: Optimized MRI of Patients With Hip Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Radiological Society of North America (Other); ISS, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-00971
Record Dates: First submitted 2021-05-04; First posted 2021-05-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Hip Arthropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MRI group (Experimental): Subjects enrolled in this study will undergo both standard and new MRI techniques. The standard MRI is needed for your routine care and as ordered by the referring doctor. The new MRI is performed for research purposes. Participants will be imaged with both methods and the results will be compared.
  Interventions: Device: Modified MRI

INTERVENTIONS:
Device: Modified MRI — A technical modification to the standard MRI which only affects radiofrequency pulse polarization attempting to optimize the image quality. All other factors, including pulse sequence parameters, and patient and coil positioning is similar to that of the standard MRI.

SUMMARY:
This is a single-center single-arm clinical trial with a paired design which compares the effectiveness of 3T MRI with (modified) and without (standard) radiofrequency pulse polarization optimization in reducing metal-related artifacts in patients with hip arthroplasty implants.

DETAILED DESCRIPTION:
Twenty participants with symptomatic primary total hip arthroplasty will be imaged with both methods. The results of the two methods will be compared in reference to the size of the artifact-degraded regions, visibility of the normal structures and the rate of abnormality detection.Primary Objective: To assess the size of the artifact-degraded regions, defined as regions of the image where underlying anatomic structure are obscured, between modified and standard MRI protocols. Secondary Objectives: (1) To assess the visibility of normal structures between modified and standard MRI protocols. (2) To assess the abnormality detection rate using modified and standard MRI protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 with unilateral symptomatic (e.g. pain) total hip arthroplasty
* Referred for MRI examination at the discretion of the treating physician
* Provision of signed and dated informed consent form
* No metal hardware in the body including contralateral hip arthroplasty
* No contraindication to MRI: defined as claustrophobia or presence of other MRI-incompatible devices

Exclusion Criteria:

* History of revision hip arthroplasty
* Pregnancy (self-reported, or self-suspected)
* Hip arthroplasty surgery within one year of enrollment
* Clinical indication to administer intravenous contrast material during MRI

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the size of the artifact-degraded regions | Visit 1, Day 0
  The area of artifact degraded regions (in pixel^2) in paired images of modified and standard MRIs determined by manual segmentation.

SECONDARY OUTCOMES:
Assessment of the visibility of normal structures | Visit 1, Day 0
  Visibility of anatomic landmarks (hip flexor, external rotator and abductor tendon attachments, joint capsule and implant-bone interface) on paired images of modified and standard MRIs using a 3-point scale with 1=structure visible without artifacts, 2=structure partly visible because of artifacts and 3=structure not visible because of artifacts
Assessment of the abnormality detection rate | Visit 1, Day 0
  Presence or absence of abnormality in paired images of modified and standard MRIs. Abnormalities include: bone marrow edema (defined as osseous short-tau inversion recovery (STIR) signal hyperintensity); fractures (linear osseous signal abnormality and osseous STIR signal hyperintensity); osteolysis (interposing linear or geographic signal hyperintensity between the host bone marrow and the implant surface); synovitis (capsular thickening and/or joint fluid with bulging of the capsule); tendinopathy (at least partial-thickness substance loss of the cross-sectional tendon area and/or split); extracapsular collections.

CONTACTS AND LOCATIONS:
Overall Officials: Iman Khodarahmi, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Radiology - Center for Biomedical Imaging, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Upon reasonable request. Requests should be directed to Iman.Khodarahmi@nyulangone.org . To gain access, data requestors will need to sign a data access agreement.